CLINICAL TRIAL: NCT07092995
Title: Leveraging Invasive Recordings and Immersive Virtual Reality to Characterize Freezing of Gait Mechanisms in Parkinson Disease
Brief Title: Understanding Freezing of Gait Using Brain Signals and Virtual Reality
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Kathryn A. Cross, MD, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-5770; 1R01NS140283 (NIH)
Record Dates: First submitted 2025-07-16; First posted 2025-07-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Parkinson&Amp;#39;s Disease; Freezing of Gait; Freezing of Gait Symptoms in Parkinson&Amp;#39;s Disease
Keywords: Deep brain stimulation; Freezing of gait; Walking; Globus pallidus internus (GPi); gait; virtual reality; electroencephalography (EEG)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Neurophysiology and kinematics are measured during gait interventions
  Interventions: Behavioral: VR Freezing Task; Behavioral: Dual Task; Behavioral: External Cueing

INTERVENTIONS:
Behavioral: VR Freezing Task — Walking overground in immersive virtual reality (VR) environments that provoke freezing episodes
Behavioral: Dual Task — Walking overground with and without concomitant performance of secondary cognitive or motor task
Behavioral: External Cueing — Walking overground in immersive virtual reality (VR) environments that provoke freezing episodes with and without addition of visual and auditory cues.

SUMMARY:
Freezing of gait - the inability to start or continue walking - is a particularly disabling problem in Parkinson's disease that has few treatment options. This project records human brain activity from deep brain stimulation (DBS) devices during walking and freezing of gait episodes to understand the pathophysiology of freezing of gait. Findings will lay the foundation for the development of new treatment strategies that address this disabling symptom.

DETAILED DESCRIPTION:
The pathophysiology of FOG is poorly understood, likely contributing to disappointing results of novel neuromodulation strategies. The goal of this study is to identify electrophysiological mechanisms of FOG that can serve as biomarkers for novel neuromodulation strategies. Activity in the globus pallidus internus (GPi), the major output nucleus of the basal ganglia, is central to understanding basal ganglia contributions to gait impairment, as it provides insights into activity that downstream locomotor circuits read out from the basal ganglia. The project leverages a state-of-the-art multimodal brain/behavior recording platform and recent advances in sensing deep brain stimulation devices to record neural activity from the human GPi simultaneously with electroencephalography (EEG), motion capture and eye gaze during over-ground walking and FOG episodes in PD patients with and without FOG. To reliably elicit FOG episodes and improve external validity, the investigators implement a novel immersive virtual reality environment to recapitulate real-world scenarios that commonly trigger FOG. With these tools, the proposed studies will determine how gait-related neural oscillations in the beta (12-30 Hz) and theta/alpha (4-12 Hz) bands in the GPi and cortex relate to abnormal gait during continuous walking (Aim 1); the onset and recovery from FOG episodes (Aim 2); and the therapeutic benefits from external cues (Aim 3). This paves the way for multiple innovative neuromodulation strategies that (1) prevent FOG episodes by promoting normal or compensatory gait control during continuous walking and (2) ameliorate severity of FOG episodes by targeting signals associated with FOG onset and recovery. Additionally, it establishes a novel VR paradigm for future precision-medicine approaches to FOG therapeutic development.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the MDS clinical diagnostic criteria for Parkinson's disease who are implanted with a Medtronic Percept DBS Device and SenSight Directional Leads in bilateral globus pallidus internus (GPi).
* Able to walk unassisted indoors
* Age 18 or older
* Half of patients will have disabling freezing of gait as defined by freezing more than once per day by self-report on questions 1 & 2 of the New Freezing of Gait Questionnaire
* The other half of patients will not have freezing of gait as defined by self-report on question 1 of the New Freezing of Gait Questionnaire

Exclusion Criteria:

* Clinical diagnosis of dementia or severe cognitive impairment (MOCA < 21)
* History of stroke, traumatic brain injury, or other neurologic disorders besides Parkinson's disease
* Comorbidities causing severe gait impairments
* Unstable medical condition including cardio-vascular instability in the past 6 months
* Unable or unwilling to comply with the testing protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
GPi gait-related spectral power | Day 1
  Globus pallidus internus (GPi) spectral power change during walking versus standing rest.
GPi event-related spectral power | Day 2
  Globus pallidus internus (GPi) spectral power changes from baseline time-locked to gait cycle events, freezing episodes, and voluntary stopping events
GPi gait-related spectral power | Day 3
  Globus pallidus internus (GPi) spectral power change during walking with versus without external cues.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share only de-identified individual-participant level (IPD) data including demographics, raw electrophysiology, timestamps from annotated video, minimally pre-processed kinematic, and eye tracking data (interpolated markers and timeseries of fixation target).
Supporting Information: Study Protocol, Analytic Code
Time Frame: At the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period.
Access Criteria: Data will be made available in the Data Archive for Brain Initiative (DABI) data repository (or equivalent), which restricts access to the data to qualified investigators with an appropriate research question and approved data use agreement (DUA) that limits subsequent use to the terms of the approved request and requires that users maintain data security, and refrain from any attempts to re-identify research participants or engage in any unauthorized uses of the data. To get access to the data, the user must submit a valid scientific question, include a statistical analysis plan, and complete all required fields on the DABI data request form. When users request access to data stored in DABI, the owners of those data are the only ones who can grant or deny access (in this case the PI).